CLINICAL TRIAL: NCT05920473
Title: Efficacy and Safety of Repetitive Transcranial Magnetic Stimulation (rTMS) for Treating Movement Disorders in Patients With Intracranial Hemorrhage (ICH): A Randomized, Blinded, Sham-controlled Trial.
Brief Title: Efficacy and Safety Study: Repetitive Transcranial Magnetic Stimulation (rTMS) for Treating Movement Disorders in Patients With Intracranial Hemorrhage (ICH).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Rehabilitation Hospital Affiliated to National Research Center for Rehabilitation Technical Aids (Unknown); Shenzhen Qianhai Shekou Free Trade Zone Hospital (Unknown)
Responsible Party: Principal Investigator, Dr. Yong Cao, director, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICH-rTMS
Record Dates: First submitted 2023-06-04; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral Hemorrhage; Movement Disorders; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cerebral Hemorrhage; Movement Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS intervention group (Experimental): Participants will undergo rTMS treatment using the Magstim Rapid 2 magnetic stimulation device. The coil was placed positioned tangentially on the scalp, targeting the hot spot (thumb movement area) in the ipsilateral cerebral hemisphere. The stimulation protocol will involve 10-Hz stimulation for 2 seconds, followed by a followed by a 10-second rest, which was repeated 50 times. Patients will receive treatment once a day, five days a week (Monday to Friday), for a total of two consecutive weeks.
  Interventions: Device: rTMS with Magstim Rapid 2 magnetic stimulation device
- Sham group (Sham Comparator): Patients in the sham group underwent sham stimulation using the Magstim Rapid 2 magnetic stimulation device with the same protocol. The coil was positioned to target the same hot spot, with an angulation parallel to the gyrus to the gyrus in order to additionally minimize the rTMS effect.
  Interventions: Device: sham control with Magstim Rapid 2 magnetic stimulation device

INTERVENTIONS:
Device: rTMS with Magstim Rapid 2 magnetic stimulation device — The study will involve the utilization of the Magstim Rapid 2 magnetic stimulation device to administer rTMS treatment to the participants. The coil will be positioned tangentially on the scalp, specifically targeting the hot spot (thumb movement area) in the ipsilateral cerebral hemisphere. During the stimulation protocol, a 10-Hz stimulation will be applied for 2 seconds, followed by a 10-second rest period. This cycle will be repeated 50 times. The treatment will be administered once daily, from Monday to Friday, for a continuous period of two weeks.
  Arms: rTMS intervention group
Device: sham control with Magstim Rapid 2 magnetic stimulation device — In the sham group, patients received sham stimulation using the the Magstim Rapid 2 magnetic stimulation device with the same protocol. The coil was positioned to target the same hot spot, with an angulation parallel to the gyrus to further reduce the potential impact of rTMS.
  Arms: Sham group

SUMMARY:
This pilot study aims to assess the effectiveness and safety of rTMS in the treatment of movement disorders in patients with ICH.

DETAILED DESCRIPTION:
While the fatality rate of intracerebral hemorrhage (ICH) has decreased, many patients continue to experience persistent limb movement dysfunction. Motor dysfunction in ICH is commonly attributed to basal ganglia hemorrhage, as the basal ganglia play a central role in the extrapyramidal motor system. Therefore, promoting the remodeling of the extrapyramidal motor system holds great significance for effectively treating ICH patients with movement disorders.

Repetitive transcranial magnetic stimulation (rTMS) is a safe and non-invasive neuromodulation technique that can modulate neuronal activity, influence neuronal synaptic plasticity, and enhance brain function. Currently, rTMS has shown promise in improving motor function among patients with stroke and those who have undergone brain tumor surgery, which provides valuable insights for its potential application in patients with motor dysfunction following ICH surgery.

This pilot study aims to evaluate the efficacy and safety of rTMS in the treatment of ICH patients with movement disorders. The participants will be randomly assigned to either a real rTMS treatment group or a sham group. The study will assess and compare various clinical outcomes, including the FMA (Fugl-Meyer Assessment), NIHSS (National Institutes of Health Stroke Scale), and BI (Barthel Index) scores, over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants between the ages of 45 and 65 years old.
2. More than 1 month and less than 3 months after ICH
3. With severe and moderately severe motor functional impairment, indicated by a Functional Motor Assessment (FMA) score ranging from 0 to 55.
4. Unilateral basal ganglia hemorrhage with a hematoma volume of 30-60ml, measured using the ABC2 method based on preoperative CT scans.
5. Participants should have a stable level of consciousness, with a score of 0 to 1 on the level of consciousness, level of consciousness questions, and level of consciousness instructions of the National Institutes of Health Stroke Scale (NIHSS), along with stable vital signs.
6. Underwent surgical treatment for ICH within 2 weeks after the event, utilizing either craniotomy or endoscopic hematoma evacuation, with an evacuation rate of at least 80%.
7. Signed the informed consent.

Exclusion Criteria:

1. With a history of epilepsy.
2. With movement disorders resulting from causes other than basal ganglia hemorrhage.
3. With severe general impairment or coexisting medical conditions.
4. With emotional issues or cognitive impairments, as indicated by a Mini-Mental State Examination (MMSE) score below 21.
5. With any contraindications to transcranial magnetic stimulation (TMS), such as having metal implants in the brain or using a pacemaker.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) | Month 6
  Motor function was evaluated using the FMA, a scale ranging from 0 to 100 that measures movement ability. Higher scores reflect better motor function. The outcome measure assesses the change in the FMA score at 6 months compared to baseline.

SECONDARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) | Day 1, Month 1, Month 3
  Motor function was evaluated using the FMA, a scale ranging from 0 to 100 that measures movement ability. Higher score reflect better motor function. The outcome measure assesses the change in the FMA score at 1 day, 1month, and 3 months compared to baseline.
Fugl-Meyer Assessment (FMA) Response | baseline, Day 1, Month 1, Month 3, Month 6
  Motor function was assessed using the FMA, which utilizes a scale ranging from 0 to 100. Higher scores indicate improved movement function, and an increase of 10 or more points in the FMA is considered a significant improvement. The response rate of the FMA was calculated at 1 day, 1 month, 3 months, and 6 months following therapy.
Change in Fugl-Meyer Assessment, Upper Limb (FMA-UL) | Day 1, Month 1, Month 3, Month 6
  Motor function of upper limb was evaluated using the FMA-UL, a scale ranging from 0 to 66 that measures upper limb movement ability. Higher score reflect better motor function. The outcome measure assesses the change in the FMA-UL score at 1 day, 1month, 3 months, and 6 months compared to baseline.
Change in Fugl-Meyer Assessment, Lower Limb (FMA-LL) | Day 1, Month 1, Month 3, Month 6
  Motor function of lower limb was evaluated using the FMA-LL, a scale ranging from 0 to 34 that measures lower limb movement ability. Higher score reflect better motor function. The outcome measure assesses the change in the FMA-LL score at 1 day, 1month, 3 months, and 6 months compared to baseline.
Change in Barthel Index (BI) score | Day 1, Month 1, Month 3, Month 6
  The activities of daily living was evaluated using the BI scores, which is a scale ranging from 0 to 100. Higher score reflect better motor function. The outcome measure assesses the change in the BI score at 1 day, 1month, 3 months, and 6 months compared to baseline.
Change in NIH stroke scale (NIHSS) score | Day 1, Month 1, Month 3, Month 6
  The stroke impairment was evaluated using the NIHSS, which is a scale ranging from 0 to 42. Higher score reflect worse function. The outcome measure assesses the change in the NIH stroke scale score at 1 day, 1month, 3 months, and 6 months compared to baseline.

OTHER OUTCOMES:
Changes in the structural brain network connectivity | Month 6
  Using Diffusion Tensor Imaging (DTI) to assess the connectivity of the brain structural network, DTI reveals the connectivity by measuring the diffusion direction and rate of water molecules in the tissue. Based on DTI, the changes in the connectivity of the brain structural network are compared between 6 months after treatment and the baseline level.
Changes in the functional brain network connectivity | Month 6
  Using functional Magnetic Resonance Imaging (fMRI) to assess the connectivity of the brain functional networks. fMRI is based on the principles of magnetic resonance and measures changes in blood oxygenation levels to reflect the activity of brain regions. Based on fMRI, the changes in connectivity of the brain functional networks are compared between 6 months after treatment and the baseline level.
Changes in the resting state brain network connectivity | Month 6
  Using resting state functional Magnetic Resonance Imaging (rs-fMRI) to assess the connectivity of the brain resting-state network. Rs-fMRI examines the changes in blood oxygenation levels in different regions during rest, revealing the state of the resting-state neural networks. Based on rs-fMRI, the changes in connectivity of brain resting-state network are compared between 6 months after treatment and the baseline level.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Cao, M.D., Principal Investigator — Department of Neurosurgery, Beijing Tiantan Hospital, Capital Medical University
Locations (3):
- China (3):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Rehabilitation Hospital Affiliated to National Research Center for Rehabilitation Technical Aids, Beijing
  - Shenzhen Qianhai Shekou Free Trade Zone Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No